CLINICAL TRIAL: NCT07048574
Title: TIDES 2.0: Prevalence and Longitudinal Course of Depression, Anxiety, and Behavior Problems in Children With Cystic Fibrosis Under 12 Years of Age
Acronym: TIDES 2
Status: Recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Brown University (Other)
Responsible Party: Principal Investigator, Beth A Smith, MD, Principal Investigator, State University of New York at Buffalo
Other Study IDs: STUDY00008868; SMITH 24A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2025-06-08; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cystic Fibrosis (CF)
Keywords: Cystic Fibrosis; Children; Mental health screening; Depression; Anxiety; CFTR modulators; Neuropsychiatric adverse events
MeSH Terms: conditions — Cystic Fibrosis; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preschool / Early Childhood Group (18 mos - 5 years): 300 children with CF and their parents will be recruited. This cohort will help identify early signs of internalizing and externalizing behaviors, attention-related concerns, and the impact of CF treatments on psychosocial health.
  Children in this cohort may also be identified for participation in Aim 3 if they are on or eligible for modulator therapy.
- School-Age Group (6 - 11 years): 300 children with CF and their parents will be recruited. Includes school-aged children who can self-report their emotional and behavioral health, beginning at age 8 years.
  This group will be assessed for emerging mental health symptoms, cognitive development, and procedural anxiety related to CF treatments.
  Children in this cohort may also be identified for participation in Aim 3 if they are on or eligible for modulator therapy.

SUMMARY:
This is a longitudinal, observational epidemiological study designed to estimate the prevalence of depression, anxiety, and behavior problems in children ages 18 months through 11 years with cystic fibrosis (CF).

DETAILED DESCRIPTION:
Integration of mental health (MH) screening and treatment into cystic fibrosis (CF) care represents over 10 years of research and clinical progress, driven by elevated rates of depression and anxiety in the International Depression Epidemiological Study, MH guidelines, and CF Foundation implementation support to screen adolescents and adults in all CF Centers. Benefits of screening include earlier identification, greater access to care, reduced stigma, and positive uptake from the CF community.

However, TIDES did not include children with CF under 12 years. Depression and anxiety have increased dramatically in young children, with new guidelines for MH screening of children in primary care. Given the pediatric MH crisis and the widespread adoption of cystic fibrosis fibrosis transmembrane conductance regulator (CFTR) modulator therapy, which have been associated with adverse events, there is an urgent need to gather MH data in children with CF <12 years. Thus, the goals of this study are to evaluate the national, longitudinal prevalence of depression, anxiety, and behavior problems in children with CF 18 months through 11 years, evaluate and compare the performance of two widely used brief screeners (criterion validity, sensitivity, specificity) to identify the optimal measures for this population, and characterize neuropsychiatric adverse events (AEs) associated with CFTR modulator therapy in this age group. Purposive randomized sampling will be used to recruit 600 children (half 18 mos.-5 yrs. and half 6-11 yrs.) at 16 CF Centers across the US. This study will estimate the prevalence of children above the clinical cut-score on each symptom domain (depression, anxiety, behavior problems) and evaluate their longitudinal course and predictors. Rigorous mixed methods will be used to describe any potential AEs perceived by parents or children to be associated with CFTR modulator therapy. This study will provide the groundwork to extend mental health screening and care to younger children with CF.

ELIGIBILITY:
Inclusion Criteria:

1. Child with a diagnosis of Cystic fibrosis (CF) actively followed by the CF care team at a participating site
2. Child is age 18 months thru 11 years
3. English and/or Spanish speaking
4. Parent/legal guardian willing and able to give informed consent, and for minor participants ages 7 thru 11 years able to give assent.

Exclusion Criteria:

* Unable or unwilling to participate in study procedures, or at Site PI discretion.

Ages: 18 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Cystic Fibrosis between 18 months and 11 years
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
To estimate the national prevalence of depression, anxiety, and behavior problems longitudinally in early childhood (18 months - 5 years) and school-age children (6 - 11 years) | 07/01/2024 - 06/30/2028
  Parents/caregivers will complete the Behavior Assessment System for Children, Third Edition (BASC-3). Children aged 8-11 years will complete the BASC-3 self-report.

SECONDARY OUTCOMES:
Evaluate and compare the performance of Pediatric Symptom Checklist (PSC) and Patient Reported Outcomes Measurement Information System (PROMIS ) compared to the Behavior Assessment System fo Children, Third Edition (BASC). | 07/01/2024 - 06/30/2028
  Parents/caregivers and children with CF will complete screening measures 3 times. The PSC and PROMIS (depression, anxiety, anger, sleep disturbance, flexibility, persistence, and cognitive function) will be assessed for sensitivity, specificity, and net benefit compared to BASC-3 clinical scales and composite indices.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Joe DiMaggio, Hollywood, Florida
  - Nemours Foundation, Orlando, Florida
  - Indiana University, Bloomington, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University at Buffalo, Buffalo, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Brown University Health, Providence, Rhode Island
  - UT Southwestern, Plano, Texas
  - Children's Hospital of Richmond at Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
An application process will be established for external data requests. Initially, data access will be granted upon request by Brown University Health (BUH), with full public access only after a defined period following study completion.
  Beyond academic publications, BUH will contribute to the creation of publicly available study summaries, ensuring that key findings are accessible to the CF community, healthcare providers, and patient advocacy groups.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Quittner AL, Goldbeck L, Abbott J, Duff A, Lambrecht P, Sole A, Tibosch MM, Bergsten Brucefors A, Yuksel H, Catastini P, Blackwell L, Barker D. Prevalence of depression and anxiety in patients with cystic fibrosis and parent caregivers: results of The International Depression Epidemiological Study across nine countries. Thorax. 2014 Dec;69(12):1090-7. doi: 10.1136/thoraxjnl-2014-205983. Epub 2014 Sep 21. PMID 25246663